CLINICAL TRIAL: NCT05889364
Title: AI-based System for Lung Tuberculosis Screening: Diagnostic Accuracy Evaluation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department (Other)
Responsible Party: Principal Investigator, Anton V. Vladzymyrskyy, Deputy CEO, Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Other Study IDs: 2018-1
Record Dates: First submitted 2018-03-28; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Tuberculosis, Pulmonary
Keywords: AI; deep learning; tuberculosis; radiology; x-ray; e-health; screening; chest; artificial intelligence
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sample N1: (n=140) with ratio "normal: tuberculosis" 50:50
  Interventions: Diagnostic Test: AI-based x-ray analysis and triage ("normal/tuberculosis suspected")
- Sample N2: (n=150) with ratio "normal: tuberculosis" 95:5
  Interventions: Diagnostic Test: AI-based x-ray analysis and triage ("normal/tuberculosis suspected")

INTERVENTIONS:
Diagnostic Test: AI-based x-ray analysis and triage ("normal/tuberculosis suspected") — All included x-rays will be analysed by the AI-based system. Then results will be compared with opinions of 2 experienced radiologists (they make peer-review of all included images independently of each other).
  Other Names: artificial intelligence analysis of medical images

SUMMARY:
Testing of AI solutions to assess diagnostic accuracy for tuberculosis detection.

DETAILED DESCRIPTION:
Tuberculosis remains a key problem of modern medicine. New approaches for burden overcoming should be proposed. New screening strategies may include artificial intelligence (AI). An AI-based system for chest x-ray analysis and triage ("normal/tuberculosis suspected") have been developed and trained. A special data-set was prepared. There are 238 normal x-rays and 70 x-rays with lung tuberculosis in data-set. The data-set was randomly divided into 2 samples:

* sample N1 (n=140) with ratio "normal: tuberculosis" 50:50,
* sample N1 (n=150) with ratio "normal: tuberculosis" 95:5. Both samples will be analysed by AI-based system. Results will be quantified using diagnostic accuracy metrics: sensitivity and specificity, positive and negative predictor values, likelihood ratio, and area under the ROC (receiver operating characteristic) curve.

ELIGIBILITY:
Inclusion Criteria:

* no pathology in a lung on chest x-ray
* signs of lung tuberculosis on chest x-ray

Exclusion Criteria:

* any pathology in the lungs (except tuberculosis)

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 308 chest x-ray images selected from the database of Unified Radiological Information Service (URIS) of Moscow
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy metric 1 | Day 1 upon receipt of data
  Sensitivity
Diagnostic accuracy metric 2 | Day 2 upon receipt of data
  Specificity
Diagnostic accuracy metric 3 | Day 3 upon receipt of data
  Positive predictor values
Diagnostic accuracy metric 4 | Day 4 upon receipt of data
  Negative predictor values
Diagnostic accuracy metric 5 | Day 5 upon receipt of data
  Likelihood ratio
Diagnostic accuracy metric 6 | Day 6 upon receipt of data
  Area under the ROC curve

CONTACTS AND LOCATIONS:
Overall Officials: Anton Vladzymyrskyy, Principal Investigator — Research and Practical Clinical Center for Diagnostics and Telemedicine Technologies of the Moscow Health Care Department
Locations (1):
- Research and Practical Center of Medical Radiology, Department of Health Care of Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No